CLINICAL TRIAL: NCT03353220
Title: Central Mechanisms and Predictors of Lorcaserin-Induced Weight Loss
Brief Title: Predictors of Lorcaserin-Induced Weight Loss
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The FDA advised of a possible health risk associated with lorcaserin and the drug is being withdrawn.
Sponsor: Columbia University (Other)
Collaborators: New York State Psychiatric Institute (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sharon Wardlaw, Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AAAR1622; 2R01DK093920 (NIH)
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Weight Loss; Lorcaserin; Healthy Volunteers
MeSH Terms: conditions — Overweight; Obesity; Weight Loss | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Participants receive lorcaserin (Belviq) 10 mg twice a day for 7 days followed by a 3 week washout period. These participants will then be crossed over to receive placebo twice a day for 7 days.
  Interventions: Drug: Belviq; Drug: Placebo
- Arm B (Experimental): Participants receive placebo twice a day for 7 days followed by a 3 week washout period. These participants will then be crossed over to receive lorcaserin (Belviq)10 mg twice a day for 7 days.
  Interventions: Drug: Belviq; Drug: Placebo

INTERVENTIONS:
Drug: Belviq — Belviq is an oral drug
  Other Names: Lorcaserin
Drug: Placebo — The placebo is made to mimic Belviq, but does not contain any active drug

SUMMARY:
This two-phase study aims to explore ways to predict who will respond well to the weight loss drug lorcaserin and to understand the mechanisms that develop which limit drug efficacy. Subjects will be recruited for a 5-week crossover study (phase 1) with lorcaserin and placebo followed by treatment with lorcaserin for 24 weeks (phase 2).

DETAILED DESCRIPTION:
In phase 1, at Weeks 1 and 5, participants will take the weight loss drug lorcaserin or placebo for 7 days. At Week 5 participants will receive whichever treatment they did not receive at Week 1. At the end of Weeks 1 and 5, participants will have a lumbar puncture (spinal tap) to collect cerebrospinal fluid (CSF) for neuropeptide and hormone analyses, including proopiomelanocortin (POMC), Agouti-related protein (AgRP) and cortisol. Blood will also be obtained for neuropeptide and hormone analyses. Breakfast will be served to participants who will then complete an eating behavior profile. A laboratory test meal will be performed 4h after breakfast.

After completing both the 7 day lorcaserin and placebo studies, participants will then continue on Phase 2 of the study, which includes treatment with lorcaserin for 24 weeks. Subjects will receive nutritional counseling to reduce their daily caloric intake to 600 kcal below their calculated caloric requirement and will be encourage to exercise moderately for 30 minutes daily. Participants will visit the clinic monthly during the 24 week study period for nutritional counseling, review of food diaries, vital signs and safely labs. Blood will also be obtained for neuropeptide peptide and hormone analyses. At the end of the 24 week period subjects will come for a final study visit, including a lumbar puncture, blood sample, breakfast, an eating behavior profile and a test meal.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 28-40

Exclusion Criteria:

* Any clinically significant or relevant medical condition, including:
* Diabetes
* Uncontrolled Hypertension
* Heart disease
* Bleeding disorder
* Kidney or liver dysfunction
* Neurologic disease
* Psychiatric or eating disorders
* Pregnancy or breastfeeding
* Use of tobacco or opiates
* History of alcohol or drug abuse
* Recent weight change +/- 5%
* Medications that affect body weight

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Wardlaw, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sideri Gugger A, Dimino C, Panigrahi SK, Mayer L, Smiley RM, Korner J, Wardlaw SL. Defining Predictors of Weight Loss Response to Lorcaserin. J Clin Endocrinol Metab. 2023 Aug 18;108(9):2262-2271. doi: 10.1210/clinem/dgad139. PMID 36897161
- See also: NIH - lorcaserin HCl — https://druginfo.nlm.nih.gov/drugportal/name/lorcaserin%20hcl
- See also: FDA approval Belviq — https://www.accessdata.fda.gov/scripts/cder/daf/index.cfm?event=overview.process&ApplNo=022529

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 32 enrolled subjects: 30 subjects completed Phase 1 (Arms A and B) and 30 subjects continued into Phase 2. However, the study was stopped prematurely during Phase 2 as lorcaserin was withdrawn from the market. Data was collected and analyzed for the 30 subjects that completed phase 1 out of 32 subjects; the 2 subjects who did not complete phase 1 were excluded from analysis. 19 subjects completed phase 2.
Groups:
- Arm A (LOR-Placebo-LOR): Phase 1: Participants receive lorcaserin (Belviq) 10 mg twice a day for 7 days followed by a 3 week washout period. These participants will then be crossed over to receive placebo twice a day for 7 days.
  Phase 2: Participants will receive additional lorcaserin (Belviq) for 24 weeks.
  Belviq: Belviq is an oral drug. Placebo: The placebo is made to mimic Belviq, but does not contain any active drug.
- Arm B (Placebo-LOR-LOR): Phase 1: Participants receive placebo twice a day for 7 days followed by a 3 week washout period. These participants will then be crossed over to receive lorcaserin (Belviq) 10 mg twice a day for 7 days.
  Phase 2: Participants will receive additional lorcaserin (Belviq) for 24 weeks.
  Belviq: Belviq is an oral drug. Placebo: The placebo is made to mimic Belviq, but does not contain any active drug.
Period: First Intervention (7 Days) - Phase 1
Arm/Group | Arm A (LOR-Placebo-LOR) | Arm B (Placebo-LOR-LOR)
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Washout (3 Weeks) - Phase 1
Arm/Group | Arm A (LOR-Placebo-LOR) | Arm B (Placebo-LOR-LOR)
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Second Intervention (7 Days) - Phase 1
Arm/Group | Arm A (LOR-Placebo-LOR) | Arm B (Placebo-LOR-LOR)
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Third Intervention (6 Months) - Phase 2
Arm/Group | Arm A (LOR-Placebo-LOR) | Arm B (Placebo-LOR-LOR)
Started | 14 | 16
Completed | 10 | 9
Not Completed | 4 | 7
Not completed — Study was stopped due to unavailable study drug supply | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Arm A+B (All Participants): Phase 1: Participants either receive lorcaserin (Belviq) 10 mg twice a day for 7 days followed by a 3 week washout period then cross over to receive placebo twice a day for 7 days (Arm A) OR receive placebo twice a day for 7 days followed by a 3 week washout period then cross over to receive lorcaserin (Belviq) 10 mg twice a day for 7 days (Arm B).
  Phase 2: Participants (from both arms) will receive additional lorcaserin (Belviq) for 24 weeks.
  Belviq: Belviq is an oral drug. Placebo: The placebo is made to mimic Belviq, but does not contain any active drug.
  Belviq: Belviq is an oral drug
  Placebo: The placebo is made to mimic Belviq, but does not contain any active drug
Arm/Group | Arm A+B (All Participants)
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Differences in Food Intake During a Laboratory Test Meal After Lorcaserin for One Week Compared to Placebo
Description: This is designed to measure food Intake (average calories consumed during test meal), in order to determine if long-term lorcaserin induced weight loss is predicted by the short-term differences in calories consumed during the test meal.
Time Frame: First test meal and follow-up test meal (approximately up to 5 weeks)
Population: The data information were collected and analyzed separately for the time period of placebo or drug exposure - i.e., comparing participants receiving placebo only OR Lorcaserin only (instead of comparing Arm A and Arm B). At one point, the same participant was exposed to either placebo OR Lorcaserin. Therefore, there are 30 analyzed for placebo only and 30 analyzed for drug only.
Measure: Mean (Standard Error); unit: kcal
Groups:
- Placebo: Phase 1: These participants either received placebo before the washout OR crossed over after washout to receive placebo twice a day for 7 days.
  Placebo: The placebo is made to mimic Belviq, but does not contain any active drug.
- Lorcaserin: Phase 1: These participants received lorcaserin (Belviq) 10 mg before the washout OR crossed over after the washout to receive lorcaserin twice a day for 7 days.
  Belviq: Belviq is an oral drug.
Arm/Group | Placebo | Lorcaserin
Number analyzed (Participants) | 30 | 30
kcal | 919.8 (118.7) | 891.9 (109.0)
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin; Test type: Other; p = 0.65, t-test, 2 sided — paired t test

2. Primary Outcome: Mean Differences in POMC Concentrations (Fmol/ml) in CSF After Lorcaserin for One Week Compared to Placebo
Description: This is designed to measure mean CSF proopiomelanocortin (POMC) concentrations (fmol/ml), in order to determine if long-term lorcaserin induced weight loss can be predicted by differences in CSF POMC concentrations.
Time Frame: Baseline, up to 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: fmol/ml
Arm/Group | Placebo | Lorcaserin
Number analyzed (Participants) | 30 | 30
fmol/ml | 256.9 (18.5) | 225.0 (15.9)
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin; Test type: Other; p = 0.0001, t-test, 2 sided — paired t test

3. Secondary Outcome: CSF Concentrations of ß-endorphin
Description: Mean differences in levels of ß-endorphin, a POMC-derived peptide, in CSF after lorcaserin for one week compared to placebo in order to determine if long-term lorcaserin induced weight loss can be predicted using short-term differences in CSF concentrations of ß-endorphin.
Time Frame: Baseline, up to 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo | Lorcaserin
Number analyzed (Participants) | 30 | 30
pg/ml | 49.07 (2.6) | 55.8 (3.2)
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin; Test type: Other; p = 0.0017, t-test, 2 sided — paired t test

4. Secondary Outcome: Mean Differences in AgRP Concentrations (pg/ml) in CSF After Lorcaserin for One Week Compared to Placebo
Description: This is designed to measure mean mean Agouti-related protein (AgRP) concentrations (pg/ml) in CSF in blood in order to determine if long-term lorcaserin induced weight loss can be predicted by short-term differences in AgRP concentrations.
Time Frame: Baseline, up to 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo | Lorcaserin
Number analyzed (Participants) | 30 | 30
pg/ml | 25.9 (3.0) | 24.2 (3.1)

5. Secondary Outcome: Mean Differences in AgRP Concentrations (Fmol/ml) in Blood After Lorcaserin for One Week Compared to Placebo
Description: This is designed to measure mean Agouti-related protein (AgRP) concentrations (fmol/ml) in blood in order to determine if long-term lorcaserin induced weight loss can be predicted by short-term differences in AgRP concentrations.
Time Frame: Baseline, up to 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo | Lorcaserin
Number analyzed (Participants) | 30 | 30
pg/ml | 78.7 (7.7) | 79.2 (7.9)

6. Secondary Outcome: Mean Differences in Cortisol Concentrations (ng/ml) in CSF After Lorcaserin for One Week Compared to Placebo
Description: This is designed to measure mean Cortisol concentrations (ng/ml) in CSF in order to determine if long-term lorcaserin induced weight loss can be predicted by short-term differences in cortisol concentrations.
Time Frame: Baseline, up to 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo | Lorcaserin
Number analyzed (Participants) | 30 | 30
pg/ml | 5.7 (0.22) | 6.08 (0.33)

7. Secondary Outcome: Insulin Level
Description: This is designed to determine effects of lorcaserin on glucose homeostasis by measuring changes in insulin levels after 1 week of lorcaserin versus placebo.
Time Frame: Changes in fasting serum insulin after 1 week of lorcaserin compared to placebo.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: µIU/ml
Arm/Group | Placebo | Lorcaserin
Number analyzed (Participants) | 30 | 30
µIU/ml | 20.1 (3.27) | 13.2 (1.16)
Statistical Analysis 1: Comparison: Placebo vs Lorcaserin; Test type: Other; p = 0.0189, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 2 years
Groups:
- LOR Time Period: Phase 1: These participants received lorcaserin (Belviq) 10 mg before the washout OR crossed over after the washout to receive lorcaserin twice a day for 7 days.
  Belviq: Belviq is an oral drug.
- Placebo Time Period: Phase 1: These participants either received placebo before the washout OR crossed over after washout to receive placebo twice a day for 7 days.
  Placebo: The placebo is made to mimic Belviq, but does not contain any active drug.
Arm/Group | LOR Time Period | Placebo Time Period
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Study was stopped prematurely during Phase 2 due to lack of drug supply.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT03353220/Prot_SAP_000.pdf